CLINICAL TRIAL: NCT02521272
Title: Hypercapnia and Gas Exchange Under the Simulated Avalanche Snow
Brief Title: Hypercapnia and Gas Exchange Under the Avalanche Snow Model (HyperAvaSM)
Acronym: HyperAvaSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Czech Technical University in Prague (Other)
Collaborators: Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: VentRes-2015-01-KR
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Accident Caused by Snow Avalanche
MeSH Terms: interventions — Respiration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- air pocket (Experimental): Breathing in the simulated avalanche snow.
  Interventions: Other: Breathing in the simulated avalanche snow.; Device: air pocket

INTERVENTIONS:
Other: Breathing in the simulated avalanche snow. — Breathing in the simulated avalanche snow with zero air pocket and one-liter air pocket.
Device: air pocket — Zero air pocket or one-liter air pocket in the snow.

SUMMARY:
The aim of the study is to investigate respiratory parameters of a person in the simulated avalanche snow and consequent use of the measured data for development of a mathematical-physical model of breathing during increasing hypercapnia in the avalanche.

DETAILED DESCRIPTION:
The study is a part of a university research project aimed at studying physiological conditions and development of breathing parameters of a person breathing in the simulated avalanche snow. Presence of an air pocket and its size play an important role in survival of victims buried in the avalanche snow. Even small air pockets facilitate breathing, yet they do not provide a significant amount of fresh air for breathing. The investigators hypothesize that the size of the air pocket significantly affects the airflow resistance and work of breathing. The aim of the study is to investigate the effect of the air pocket volume on gas exchange and work of breathing in subjects breathing into the simulated avalanche snow and to test, whether it is possible to breathe with zero air pocket.

ELIGIBILITY:
Inclusion Criteria:

* Participants were volunteers from the Czech Army forces, studying at the Military Department of the Faculty of Physical Education and Sport, Charles University in Prague. All subjects were healthy and fit, classified as ASA I, all without a smoking history. The volunteers were highly motivated to participate in the experiment. The entrance examination, completed before the start of the study, included these tests: electrocardiography, blood pressure, spirometry, and assessment of the health conditions and family anamnesis by a physician with a specialty in anesthesia and critical care.

Exclusion Criteria:

* The exclusion criteria were Tiffeneau Index less than 0.70 and any cardiovascular or respiratory condition.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The length of breathing | Continuously within 30 minute interval from the beginning of the breathing experiment
  Time to termination of the breathing experiment due to the decision of the subject, or determined by high End-Tidal CO2 value or by the order by the clinician assessing the health status of the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Karel Roubik, prof., Ph.D., Study Director — Czech Technical University in Prague
Locations (1):
- Charles University, Czech Republic, Prague, Czechia

REFERENCES:
- [Background] Brugger H, Sumann G, Meister R, Adler-Kastner L, Mair P, Gunga HC, Schobersberger W, Falk M. Hypoxia and hypercapnia during respiration into an artificial air pocket in snow: implications for avalanche survival. Resuscitation. 2003 Jul;58(1):81-8. doi: 10.1016/s0300-9572(03)00113-8. PMID 12867313
- [Background] Bellani G, Patroniti N, Weismann D, Galbiati L, Curto F, Foti G, Pesenti A. Measurement of pressure-time product during spontaneous assisted breathing by rapid interrupter technique. Anesthesiology. 2007 Mar;106(3):484-90. doi: 10.1097/00000542-200703000-00012. PMID 17325506
- [Background] Grissom CK, Radwin MI, Harmston CH, Hirshberg EL, Crowley TJ. Respiration during snow burial using an artificial air pocket. JAMA. 2000 May 3;283(17):2266-71. doi: 10.1001/jama.283.17.2266. PMID 10807386